CLINICAL TRIAL: NCT03829449
Title: CONSERVE: rVA576 (Coversin) Long Term Safety and Efficacy Surveillance Study
Brief Title: rVA576 (Coversin) Long Term Safety and Efficacy Surveillance Study
Acronym: CONSERVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The early termination of this study is a business decision, Akari have made the decision to close their global Phase III PNH program. The decision was not related to any efficacy, safety or clinical concerns regarding Coversin/rVA576.
Sponsor: AKARI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK581
Record Dates: First submitted 2018-12-20; First posted 2019-02-04 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Intervention Model Description: Open-label, non-comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- rVA576 Coversin (Experimental): The study population will consist of patients who have completed participation in clinical trials under other Akari protocols and who wish to continue to receive rVA576 (Coversin) for up to 4 years.
  Interventions: Drug: rVA576

INTERVENTIONS:
Drug: rVA576 — The study population will consist of patients who have completed participation in clinical trials under other Akari protocols and who wish to continue to receive rVA576 (Coversin).
  Other Names: nomacopan

SUMMARY:
Long term management of patients with complement related diseases including Paroxysmal Nocturnal Haemoglobinuria and Atypical Haemolytic Uraemic Syndrome

DETAILED DESCRIPTION:
Patients with diseases requiring complement inhibition who have previously taken part in Akari clinical trials and who wish to continue to receive rVA576 (Coversin) after their active participation in the parent trial has completed and patients treated under compassionate use or named patient arrangements who wish to continue on rVA576 (Coversin) therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and above treated with rVA576 (Coversin) under other Akari clinical trial protocols and wish to remain on rVA576 (Coversin) at the conclusion of that trial.
2. In the opinion of the treating responsible clinician patient is receiving clinical benefit from continued treatment with study drug.
3. Evidence of sustained complement inhibition by CH50 assay. .
4. Women of childbearing potential (WOCBP) must agree to use effective contraception consistently throughout the study and have a negative pregnancy test at screening and a negative urine pregnancy test per the schedule of visits. Women cannot donate their eggs. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of amenorrhea or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks previously.
5. Males with a childbearing potential partner must agree to use effective contraception consistently OR have had a vasectomy
6. Weight ≥50-100kg
7. Willing to receive appropriate prophylaxis against Neisseria meningitidis infection, by both immunisation and continuous or intermittent antibiotics
8. The patient is willing to give voluntary written informed consent
9. The patient is willing in the process of preparation and self-administration of the study drug.

Exclusion Criteria:

1. Patient experienced any safety event in the previous study protocol, which puts the patient at unacceptable risk in current protocol as judged by the investigator and sponsor.
2. Patient is unwilling to complete the Quality of Life instruments and diary card
3. Active meningococcal infection (section 4.3.1 for additional information)
4. Any other reason for which, in the opinion of the Investigator, it would not be in the interests of the patient to remain on rVA576 (Coversin).
5. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 90 days after last dose; or intending to donate ova during such time period.
6. If male, the subject intends to donate sperm while on the study this study or for 90 days after last dose.
7. Failure to satisfy the Investigator of fitness to participate for any other reason or any other condition which, in the opinion of the investigator, could increase the subject's risk by participating in the study or confound the outcome of the study.
8. Use of prohibited medication
9. The subject has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse.
10. Participation in other clinical trials with investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wynne Weston Davies, Study Director — AKARI Therapeutics
Locations (1):
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rVA576 Coversin
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The primary analysis was intention to treat (ITT) and all patients who entered and who signed the ICF were included in the Full Analysis Set.
Groups:
- rVA576 Coversin: The study population will consist of patients who have completed participation in clinical trials under other Akari protocols and who wish to continue to receive rVA576 for up to 4 years.
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 39 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 1
  Netherlands | 1
  Poland | 5
  United Kingdom | 2
  Lithuania | 2
  Sri Lanka | 4

OUTCOME MEASURES:

1. Primary Outcome: Long Term Safety and Efficacy of rVA576 (Coversin) Therapy Assessed by AEs, SAEs, Standard Lab Tests and ECG Results.
Description: To determine the safety profile of long-term rVA576 (Coversin) treatment as assessed by AEs, SAEs, Standard Lab tests and ECG results.
Time Frame: On entry and every 3 months thereafter, for the duration of the study (approximately 3 years and 5 months)
Measure: Count of Participants; unit: Participants
Groups:
- rVA576: rVA576: The study population will consist of patients who have completed participation in clinical trials under other sponsor protocols and who wish to continue to receive rVA576 in open label single arm
Arm/Group | rVA576
Number analyzed (Participants) | 15
Participants
  Adverse Events | 14
  Serious Adverse Events | 3
  Clinically significant hemoglobin (low) | 7
  Clinically significant hematocrit (low) | 6
  Clinically significant MCH (high) | 4
  Clinically significant MCV (high) | 3
  Clinically significant RBC (low) | 6
  Clinically significant reticulocytes (high) | 4
  Clinically significant basophils (low) | 1
  Clinically significant eosinophils (low) | 1
  Clinically significant neutrophils (low) | 1
  Clinically significant platelets (low) | 1
  Clinically significant reticulocytes (low) | 2
  Clinically significant WBC (low) | 1
  Clinically significant ALT (high) | 3
  Clinically significant AST (high) | 6
  Clinically significant creatine kinase (high) | 2
  Clinically significant creatinine (high) | 6
  Clinically significant direct bilirubin (high) | 5
  Clinically significant total bilirubin (high) | 7
  Clinically significant gamma glutamyl transpeptidase (GGT) (high) | 2
  Clinically significant LDH (high) | 10
  Clinically significant potassium (high) | 1
  Clinically significant urea (high) | 2
  Clinically significant potassium (low) | 1
  Clinically significant ECG | 1

2. Secondary Outcome: Proportion of Subjects With Thrombotic and Haemolytic Event Free Status During Each 3month Time Period Since the Start of the Study.
Description: Thrombotic and Haemolytic Events will include, but are not limited to, the following: haemolytic anaemia, thrombocytopenia, red blood cell haemolysis indicated by dark urine, Budd-Chiara syndrome, any other thrombotic or haemolytic event deemed to be associated with PNH. A haemolytic event will be defined as a rise in LDH or other biochemical evidence of haemolysis accompanied by an increase in symptoms and/or frank haemoglobinuria. Increased symptoms without objective haematological or biochemical evidence of haemolysis will not be counted as haemolytic events. In addition, the following signs and symptoms may be reviewed and classified as Thrombotic/Haemolytic events if appropriate: Acute kidney failure, Hypertension, Myocardial infarction, Stroke, Lung complications, Seizure, Coma, Premature death.
Time Frame: On entry and every 3 months thereafter, for the duration of the study (approximately 3 years and 5 months)
Population: Data are not available for all 15 participants at every 3-month interval due to the early termination of the trial. The proportion of subjects with thrombotic or haemolytic event free status in each 3-month interval is calculated based on the actual number of participants analysed at each 3-month interval.
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576
Number analyzed (Participants) | 15
Participants
  Proportion of subjects with thrombotic event free status: 0 - 3 Months | 15
  Proportion of subjects with thrombotic event free status: >3 - 6 Months | 15
  Proportion of subjects with thrombotic event free status: >6 - 9 Months: number analyzed (Participants) | 11
  Proportion of subjects with thrombotic event free status: >6 - 9 Months | 11
  Proportion of subjects with thrombotic event free status: >9 - 12 Months: number analyzed (Participants) | 10
  Proportion of subjects with thrombotic event free status: >9 - 12 Months | 10
  Proportion of subjects with thrombotic event free status: >12 - 15 Months: number analyzed (Participants) | 10
  Proportion of subjects with thrombotic event free status: >12 - 15 Months | 10
  Proportion of subjects with thrombotic event free status: >15 - 18 Months: number analyzed (Participants) | 10
  Proportion of subjects with thrombotic event free status: >15 - 18 Months | 10
  Proportion of subjects with thrombotic event free status: >18 - 21 Months: number analyzed (Participants) | 8
  Proportion of subjects with thrombotic event free status: >18 - 21 Months | 8
  Proportion of subjects with thrombotic event free status: >21 - 24 Months: number analyzed (Participants) | 7
  Proportion of subjects with thrombotic event free status: >21 - 24 Months | 7
  Proportion of subjects with thrombotic event free status: >24 - 27 Months: number analyzed (Participants) | 6
  Proportion of subjects with thrombotic event free status: >24 - 27 Months | 6
  Proportion of subjects with thrombotic event free status: >27 - 30 Months: number analyzed (Participants) | 6
  Proportion of subjects with thrombotic event free status: >27 - 30 Months | 6
  Proportion of subjects with thrombotic event free status: >30 Months: number analyzed (Participants) | 5
  Proportion of subjects with thrombotic event free status: >30 Months | 5
  Proportion of subjects with haemolytic event free status: 0 - 3 Months | 13
  Proportion of subjects with haemolytic event free status: >3 - 6 Months | 11
  Proportion of subjects with haemolytic event free status: >6 - 9 Months: number analyzed (Participants) | 11
  Proportion of subjects with haemolytic event free status: >6 - 9 Months | 9
  Proportion of subjects with haemolytic event free status: >9 - 12 Months: number analyzed (Participants) | 10
  Proportion of subjects with haemolytic event free status: >9 - 12 Months | 9
  Proportion of subjects with haemolytic event free status: >12 - 15 Months: number analyzed (Participants) | 10
  Proportion of subjects with haemolytic event free status: >12 - 15 Months | 10
  Proportion of subjects with haemolytic event free status: >15 - 18 Months: number analyzed (Participants) | 10
  Proportion of subjects with haemolytic event free status: >15 - 18 Months | 10
  Proportion of subjects with haemolytic event free status: >18 - 21 Months: number analyzed (Participants) | 8
  Proportion of subjects with haemolytic event free status: >18 - 21 Months | 8
  Proportion of subjects with haemolytic event free status: >21 - 24 Months: number analyzed (Participants) | 7
  Proportion of subjects with haemolytic event free status: >21 - 24 Months | 7
  Proportion of subjects with haemolytic event free status: >24 - 27 Months: number analyzed (Participants) | 6
  Proportion of subjects with haemolytic event free status: >24 - 27 Months | 6
  Proportion of subjects with haemolytic event free status: >27 - 30 Months: number analyzed (Participants) | 6
  Proportion of subjects with haemolytic event free status: >27 - 30 Months | 6
  Proportion of subjects with haemolytic event free status: >30 Months: number analyzed (Participants) | 5
  Proportion of subjects with haemolytic event free status: >30 Months | 5

3. Secondary Outcome: Time to Thrombotic or Haemolytic Event Since Joining This Study.
Description: Time to thrombotic or haemolytic event since joining this study.
Time Frame: Approximately 3 years and 5 months
Measure: Mean (Standard Deviation); unit: days since first dose
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 14
days since first dose | 113.0 (80.61)

4. Secondary Outcome: Proportion of Subjects Who Require PRBC Transfusion During Each 3-month Period Since the Start of the Study and Over the Entire Period of the Study
Description: Proportion of subjects who require PRBC transfusion during each 3-month period since the start of the study and over the entire period of the study
Time Frame: On entry and every 3 months thereafter, for the duration of the study (approximately 3 years and 5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 15
Participants
  0 - 3 Months | 3
  >3 - 6 Months | 2
  >6 - 9 Months | 2
  >9 - 12 Months | 3
  >12 - 15 Months | 3
  >15 - 18 Months | 0
  >18 - 21 Months | 0
  >21 - 24 Months | 1
  >24 - 27 Months | 1
  >27 - 30 Months | 1
  >30 Months | 0
  Entire Study | 4

5. Secondary Outcome: Time to First Transfusion Since Joining the Study.
Description: Time to first transfusion since joining the study.
Time Frame: approximately 3 years and 5 months
Measure: Median (Full Range); unit: days
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 15
days | 30.5 [1 to 284]

6. Secondary Outcome: Proportion of Subjects With no Adverse Change in Overall Scores of Quality of Life Using the EORTC QLQ-C30, the EQ-5D-5L and FACIT-F Instruments at Each 3-month Time Period Since the Start of the Study.
Description: Proportion of subjects with no adverse change in overall scores of Quality of Life using the EORTC QLQ-C30, the EQ-5D-5L and FACIT-F instruments at each 3-month time period since the start of the study.
Time Frame: Every 3 months up to 39 months
Population: Not all participants completed the self-reported questionnaires at all timepoints
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 15
Participants
  0 - 3 Months - EORTC QLQ-C30: number analyzed (Participants) | 11
  0 - 3 Months - EORTC QLQ-C30 | 9
  >3 - 6 Months - EORTC QLQ-C30: number analyzed (Participants) | 11
  >3 - 6 Months - EORTC QLQ-C30 | 8
  >6 - 9 Months - EORTC QLQ-C30: number analyzed (Participants) | 10
  >6 - 9 Months - EORTC QLQ-C30 | 9
  >9 - 12 Months - EORTC QLQ-C30: number analyzed (Participants) | 10
  >9 - 12 Months - EORTC QLQ-C30 | 6
  >12 - 15 Months - EORTC QLQ-C30: number analyzed (Participants) | 1
  >12 - 15 Months - EORTC QLQ-C30 | 0
  >15 - 18 Months - EORTC QLQ-C30: number analyzed (Participants) | 8
  >15 - 18 Months - EORTC QLQ-C30 | 4
  >18 - 21 Months - EORTC QLQ-C30: number analyzed (Participants) | 4
  >18 - 21 Months - EORTC QLQ-C30 | 2
  >21 - 24 Months - EORTC QLQ-C30: number analyzed (Participants) | 6
  >21 - 24 Months - EORTC QLQ-C30 | 5
  >24 - 27 Months - EORTC QLQ-C30: number analyzed (Participants) | 4
  >24 - 27 Months - EORTC QLQ-C30 | 3
  >27 - 30 Months - EORTC QLQ-C30: number analyzed (Participants) | 5
  >27 - 30 Months - EORTC QLQ-C30 | 4
  >30 - 33 Months - EORTC QLQ-C30: number analyzed (Participants) | 2
  >30 - 33 Months - EORTC QLQ-C30 | 2
  >33 - 36 Months - EORTC QLQ-C30: number analyzed (Participants) | 2
  >33 - 36 Months - EORTC QLQ-C30 | 1
  >36 - 39 Months - EORTC QLQ-C30: number analyzed (Participants) | 2
  >36 - 39 Months - EORTC QLQ-C30 | 2
  0 - 3 Months - EQ-5D-5L: number analyzed (Participants) | 9
  0 - 3 Months - EQ-5D-5L | 7
  >3 - 6 Months - EQ-5D-5L: number analyzed (Participants) | 9
  >3 - 6 Months - EQ-5D-5L | 6
  >6 - 9 Months - EQ-5D-5L: number analyzed (Participants) | 9
  >6 - 9 Months - EQ-5D-5L | 8
  >9 - 12 Months - EQ-5D-5L: number analyzed (Participants) | 9
  >9 - 12 Months - EQ-5D-5L | 4
  >12 - 15 Months - EQ-5D-5L: number analyzed (Participants) | 1
  >12 - 15 Months - EQ-5D-5L | 1
  >15 - 18 Months - EQ-5D-5L: number analyzed (Participants) | 8
  >15 - 18 Months - EQ-5D-5L | 5
  >18 - 21 Months - EQ-5D-5L: number analyzed (Participants) | 4
  >18 - 21 Months - EQ-5D-5L | 2
  >21 - 24 Months - EQ-5D-5L: number analyzed (Participants) | 6
  >21 - 24 Months - EQ-5D-5L | 2
  >24 - 27 Months - EQ-5D-5L: number analyzed (Participants) | 4
  >24 - 27 Months - EQ-5D-5L | 3
  >27 - 30 Months - EQ-5D-5L: number analyzed (Participants) | 5
  >27 - 30 Months - EQ-5D-5L | 3
  >30 - 33 Months - EQ-5D-5L: number analyzed (Participants) | 2
  >30 - 33 Months - EQ-5D-5L | 2
  >33 - 36 Months - EQ-5D-5L: number analyzed (Participants) | 2
  >33 - 36 Months - EQ-5D-5L | 2
  >36 - 39 Months - EQ-5D-5L: number analyzed (Participants) | 2
  >36 - 39 Months - EQ-5D-5L | 2
  0 - 3 Months - FACIT-F: number analyzed (Participants) | 3
  0 - 3 Months - FACIT-F | 0
  >3 - 6 Months - FACIT-F: number analyzed (Participants) | 2
  >3 - 6 Months - FACIT-F | 1
  >6 - 9 Months - FACIT-F: number analyzed (Participants) | 1
  >6 - 9 Months - FACIT-F | 0
  >9 - 12 Months - FACIT-F: number analyzed (Participants) | 1
  >9 - 12 Months - FACIT-F | 0
  >12 - 15 Months - FACIT-F: number analyzed (Participants) | 0
  >12 - 15 Months - FACIT-F | 0
  >15 - 18 Months - FACIT-F: number analyzed (Participants) | 0
  >15 - 18 Months - FACIT-F | 0
  >18 - 21 Months - FACIT-F: number analyzed (Participants) | 0
  >18 - 21 Months - FACIT-F | 0
  >21 - 24 Months - FACIT-F: number analyzed (Participants) | 0
  >21 - 24 Months - FACIT-F | 0
  >24 - 27 Months - FACIT-F: number analyzed (Participants) | 0
  >24 - 27 Months - FACIT-F | 0
  >27 - 30 Months - FACIT-F: number analyzed (Participants) | 0
  >27 - 30 Months - FACIT-F | 0
  >30 - 33 Months - FACIT-F: number analyzed (Participants) | 0
  >30 - 33 Months - FACIT-F | 0
  >33 - 36 Months - FACIT-F: number analyzed (Participants) | 0
  >33 - 36 Months - FACIT-F | 0
  >36 - 39 Months - FACIT-F: number analyzed (Participants) | 0
  >36 - 39 Months - FACIT-F | 0

7. Secondary Outcome: Proportion of Subjects With Serum Lactate Dehydrogenase (LDH) <1.8, >1.8 to 2.4, >2.4 to 3, and >3 Times the Upper Limit of Normal (ULN) at Each 3-month Time Period Since the Start of the Study.
Description: Proportion of subjects with serum Lactate Dehydrogenase (LDH) <1.8, >1.8 to 2.4, >2.4 to 3, and >3 times the upper limit of normal (ULN) at each 3-month time period since the start of the study.
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | rVA576
Number analyzed (Participants) | 15
Participants | 3

8. Secondary Outcome: Proportion of Subjects With Median Serum Lactate Dehydrogenase (LDH) <1.8, >1.8 to 2.4, >2.4 to 3, and >3 Times the Upper Limit of Normal (ULN) Over the Entire Duration of the Study.
Description: Proportion of subjects with median serum Lactate Dehydrogenase (LDH) <1.8, >1.8 to 2.4, >2.4 to 3, and >3 times the upper limit of normal (ULN) over the entire duration of the study.
Time Frame: Approximately 3 years and 5 months
Measure: Number; unit: Participants
Arm/Group | rVA576
Number analyzed (Participants) | 15
Participants | 4

9. Secondary Outcome: Proportion of Transfusion-independent Subjects at Each 3-month Time Point, With Haemoglobin (g/L) Above the Baseline Haemoglobin Value They Had at the Start of the Trial From Which They Entered CONSERVE
Description: Proportion of transfusion-independent subjects at each 3-month time point, with haemoglobin (g/L) above the baseline haemoglobin value they had at the start of the trial from which they entered CONSERVE
Time Frame: Baseline and every 3 months up to 39 months
Population: Total number of subjects analyzed at each timepoint is specified.
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 11
Participants
  Baseline | 11
  Month 3: number analyzed (Participants) | 9
  Month 3 | 4
  Month 6: number analyzed (Participants) | 8
  Month 6 | 4
  Month 9: number analyzed (Participants) | 7
  Month 9 | 3
  Month 12: number analyzed (Participants) | 7
  Month 12 | 4
  Month 15: number analyzed (Participants) | 1
  Month 15 | 0
  Month 18: number analyzed (Participants) | 5
  Month 18 | 3
  Month 21: number analyzed (Participants) | 2
  Month 21 | 1
  Month 24: number analyzed (Participants) | 4
  Month 24 | 3
  Month 27: number analyzed (Participants) | 2
  Month 27 | 1
  Month 30: number analyzed (Participants) | 3
  Month 30 | 3
  Month 33: number analyzed (Participants) | 2
  Month 33 | 1
  Month 36: number analyzed (Participants) | 2
  Month 36 | 1
  Month 39: number analyzed (Participants) | 2
  Month 39 | 1

10. Secondary Outcome: Proportion of Transfusion-independent Subjects Over the Entire Duration of the Study With Mean Haemoglobin (g/L) Above the Baseline Haemoglobin Value They Had at the Start of the Trial From Which They Entered CONSERVE
Description: Proportion of transfusion-independent subjects over the entire duration of the study with mean haemoglobin (g/L) above the baseline haemoglobin value they had at the start of the trial from which they entered CONSERVE
Time Frame: Approximately 3 years and 5 months
Population: Total number of subjects analyzed with post-baseline values is specified.
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 11
Participants
  Baseline | 11
  Overall Post-Baseline Mean Haemoglobin: number analyzed (Participants) | 9
  Overall Post-Baseline Mean Haemoglobin | 4

11. Secondary Outcome: Proportion of Patients Experiencing Major Adverse Vascular Events (MAVE) Over the Entire Period of the Study.
Description: Proportion of patients experiencing Major Adverse Vascular Events (MAVE) over the entire period of the study.
Time Frame: Approximately 3 years and 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 15
Participants | 0

12. Secondary Outcome: Time to First Major Adverse Vascular Event (MAVE) for Each Subject Since Joining the Study.
Description: Time to first Major Adverse Vascular Event (MAVE) for each subject since joining the study.
Time Frame: Approximately 3 years and 5 months
Population: There were no Major Adverse Vascular Events (MAVEs) reported during the entire period of the study.
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Major Adverse Vascular Events (MAVE) Over the Entire Period of the Study.
Description: Number of Major Adverse Vascular Events (MAVE) over the entire period of the study.
Time Frame: Approximately 3 years and 5 months
Measure: Number; unit: events
Arm/Group | rVA576 Coversin
Number analyzed (Participants) | 15
events | 0

ADVERSE EVENTS:
Time Frame: Approximately 3 years and 5 months
Arm/Group | rVA576 Coversin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rVA576 Coversin (N=15)
Urinary tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Pyrexia (General disorders) | 1 (1) — System Organ Class: General disorders & administration site conditions
Intravascular haemolysis (Blood and lymphatic system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rVA576 Coversin (N=15)
Urinary tract infection (Infections and infestations) | 5 (8)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (4)
Nasopharyngitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 3 (8)
Renal failure (Renal and urinary disorders) | 2 (3)
Haemoglobinuria (Renal and urinary disorders) | 2 (5)
Chromaturia (Renal and urinary disorders) | 2 (5)
Dysuria (Renal and urinary disorders) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 4 (5) — System Organ Class: General disorders & administration site conditions
Influenza like illness (General disorders) | 1 (3) — System Organ Class: General disorders & administration site conditions
Fatigue (General disorders) | 2 (2) — System Organ Class: General disorders & administration site conditions
Injection site pain (General disorders) | 1 (2) — System Organ Class: General disorders & administration site conditions
Injection site pruritus (General disorders) | 1 (1) — System Organ Class: General disorders & administration site conditions
Injection site swelling (General disorders) | 1 (1) — System Organ Class: General disorders & administration site conditions
Urinary casts (Investigations) | 2 (2)
White blood cells urine positive (Investigations) | 2 (2)
Blood LDH increased (Investigations) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1)
WBC decreased (Investigations) | 1 (1)
Glucose urine present (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the early termination of this study, only a subset of the outputs planned were produced. Parent trial locked databases were not pooled with the AK581 database, limiting the scope of the analyses that could be produced. The 'parent trial baseline' could not be used in calculations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03829449/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03829449/SAP_001.pdf